CLINICAL TRIAL: NCT01149278
Title: Assessment of Two Levels of Arterial Pressure on Survival in Patients With Septic Shock
Acronym: SEPSISPAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Pr ASFAR Pierre, University Hospital, Angers
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC09-01
Record Dates: First submitted 2010-06-09; First posted 2010-06-23 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2010-06

CONDITIONS: Septic Shock; Arterial Pressure; Hemodynamics; Mortality; Clinical Trial
MeSH Terms: conditions — Shock, Septic

ARMS (2):
- high pressure (Active Comparator)
  Interventions: Drug: maintain mean arterial pressure between 80-85 mm Hg
- normal pressure (Placebo Comparator)
  Interventions: Other: maintain mean arterial pressure between 65-70 mm Hg

INTERVENTIONS:
Drug: maintain mean arterial pressure between 80-85 mm Hg — protocolized hemodynamic care aiming to maintain mean arterial pressure between 80-85 mm Hg
  Arms: high pressure
Other: maintain mean arterial pressure between 65-70 mm Hg — protocolized hemodynamic care aiming to maintain mean arterial pressure between 65-70 mm Hg
  Arms: normal pressure

SUMMARY:
The ideal mean arterial pressure in patients with septic shock is unknown. The expert's recommandations have stated a target between 65 and 70 mm Hg. However the scientific basis are weak. Indead there are only few prospective studies which addressed this question without clear answer. Therefore we designed a RCT in order to assess the effect on mortality of two levels of mean arterial pressure in patients with septic shock.(800 patients, 30 centres)

ELIGIBILITY:
Inclusion Criteria:

* patients with septic shock according criteria of Bone
* minimal dose of norepinephrine
* Written informed consent obtained from the patient or surrogate

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Participation in other trials with the same endpoints
* moribund
* absence of registration in french health care system
* patient protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2010-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
mortality | day 28

SECONDARY OUTCOMES:
decrease in mortality at day 90 | day 90
decrease in sequential organ failure assessment | day 1 to day 28
extra renal replacement free days | day 28
renal function | day 1 to day 28
amount of fluids | day 1 to end of shock
catecholamines free days | day 1 to day 28

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital Angers, Angers, France

REFERENCES:
- [Derived] Pirracchio R, Fong N, Legrand M. Heterogeneity in the response to a high vs low mean arterial pressure target in patients with septic shock a post hoc analysis of a randomized controlled trial. Intensive Care Med. 2025 Oct;51(10):1775-1783. doi: 10.1007/s00134-025-08104-8. Epub 2025 Sep 17. PMID 40960603
- [Derived] Asfar P, Meziani F, Hamel JF, Grelon F, Megarbane B, Anguel N, Mira JP, Dequin PF, Gergaud S, Weiss N, Legay F, Le Tulzo Y, Conrad M, Robert R, Gonzalez F, Guitton C, Tamion F, Tonnelier JM, Guezennec P, Van Der Linden T, Vieillard-Baron A, Mariotte E, Pradel G, Lesieur O, Ricard JD, Herve F, du Cheyron D, Guerin C, Mercat A, Teboul JL, Radermacher P; SEPSISPAM Investigators. High versus low blood-pressure target in patients with septic shock. N Engl J Med. 2014 Apr 24;370(17):1583-93. doi: 10.1056/NEJMoa1312173. Epub 2014 Mar 18. PMID 24635770